CLINICAL TRIAL: NCT04062552
Title: Implementing Palliative Care: Learning Collaborative vs. Technical Assistance
Brief Title: Learning Collaborative Versus Technical Assistance in Delivering a Palliative Care Program to Patients With Advanced Cancer and Their Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester NCORP Research Base (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Supriya Mohile, URCC Study Co-Chair, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: URCC18110CD; NCI-2019-02246 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC18110CD_; URCC18110CD (Other: University of Rochester NCORP Research Base); URCC-18110CD (Other: DCP); URCC-18110CD (Other: CTEP); R01CA229197 (NIH); UG1CA189961 (NIH)
Record Dates: First submitted 2019-08-12; First posted 2019-08-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Early Intervention, Educational; Educational Status; Methods; Restraint, Physical; Nutrition Surveys; Independent Medical Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (ENABLE palliative care program, phone calls, VLC) (Experimental): Patients undergo a palliative care assessment, participate in 6 ENABLE phone-based sessions with an ENABLE coach over 20-40 minutes, and monthly follow-up calls for 6 months. Caregivers participate in 3 ENABLE sessions with an ENABLE coach and monthly follow-up calls for 6 months. The practice sites participate in a VLC consisting of group-based learning sessions, coaching, and applied quality improvement data collection, analysis and feedback opportunities monthly for 15 months.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Other: Educational Intervention; Procedure: Medical Examination Assessment; Other: Quality-of-Life Assessment; Other: Survey Administration; Behavioral: Telephone-Based Intervention
- Group II (ENABLE palliative care program, phone calls, TA) (Experimental): Patients undergo a palliative care assessment, participate in 6 ENABLE phone-based sessions with an ENABLE coach over 20-40 minutes, and monthly follow-up calls for 6 months. Caregivers participate in 3 ENABLE sessions with an ENABLE coach and monthly follow-up calls for 6 months. The practice sites undergo practice-based consultation calls with an ENABLE/TA expert monthly for 15 months.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Other: Educational Intervention; Procedure: Medical Examination Assessment; Other: Quality-of-Life Assessment; Other: Survey Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Behavioral, Psychological or Informational Intervention — Receive ENABLE palliative care information
Other: Educational Intervention — Participate in VLC group-based learning sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (ENABLE palliative care program, phone calls, VLC)
Other: Educational Intervention — Participate in consultation with ENABLE/TA expert
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group II (ENABLE palliative care program, phone calls, TA)
Procedure: Medical Examination Assessment — Undergo palliative care assessment
  Other Names: Exam; Examination; Health Assessment; Health Examination; Health Status Assessment; Medical Assessment; Medical Exam; Medical Inspection
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Complete surveys
Behavioral: Telephone-Based Intervention — Receive monthly phone calls

SUMMARY:
This trial studies the delivery of the ENABLE palliative care program by two different methods called a Virtual Learning Collaborative or Technical Assistance for patients with advanced cancer and their caregivers. Palliative care is specialized medical care for people with a serious illness that occurs at the same time as other medical treatment. The purpose of palliative care is to provide relief from symptoms and stress of serious illness, to help patients and their families clarify goals of care, and to focus on social support and spiritual well-being. The focus of the ENABLE palliative care program is on living well, managing stress, patient communication of their personal values and hopes for care, social support, and symptom management. This study may help doctors find the best ways to include palliative care services into their practices and the impact of palliative care on cancer patients and their caregivers' quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Gather preliminary data on the effectiveness of virtual learning collaborative (VLC) versus (vs.) technical assistance (TA) on educate, nurture, advise before life ends (ENABLE) program uptake, defined as the proportion of patients that complete a palliative care assessment and at least 4 ENABLE sessions.

SECONDARY OBJECTIVE:

I. Evaluate the preliminary effectiveness of VLC or TA on patient quality of life (QOL) and mood outcomes.

II. Evaluate the relationship between ENABLE program uptake and patients' QOL and mood across the two strategies.

EXPLORATORY OBJECTIVES:

I. Evaluate the effectiveness of VLC vs. TA on participating institutions' overall ENABLE program implementation, as measured by the General Organizational Index (GOI).

II. Evaluate the relationship between overall ENABLE program implementation and patients' QOL and mood across the two strategies.

OUTLINE: Health care practice sites are randomized to 1 of 2 groups.

GROUP I: Patients undergo a palliative care assessment, participate in 6 ENABLE phone-based sessions with an ENABLE coach over 20-40 minutes, and monthly follow-up calls for 6 months. Caregivers participate in 3 ENABLE sessions with an ENABLE coach and monthly follow-up calls for 6 months. The practice sites participate in a Virtual Learning Collaborative (VLC) consisting of group-based learning sessions, coaching, and applied quality improvement data collection, analysis and feedback opportunities monthly for 15 months.

GROUP II: Patients undergo a palliative care assessment, participate in 6 ENABLE phone-based sessions with an ENABLE coach over 20-40 minutes, and monthly follow-up calls for 6 months. Caregivers participate in 3 ENABLE sessions with an ENABLE coach and monthly follow-up calls for 6 months. The practice sites undergo practice-based consultation calls with an ENABLE/Technical Assistance (TA) expert monthly for 15 months.

After completion of the study, participants are followed up at 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PRACTICE SITE: All participating practice clusters will be asked to identify one (or more) ENABLE coach as part of study eligibility to deliver the ENABLE program.
* PRACTICE SITE: Commitment of the ENABLE coach(es) to be trained to conduct the palliative care assessment (and ENABLE sessions if the practice plans to implement them).
* PRACTICE SITE: Desire to implement ENABLE, including presence of an investigator (e.g., primary affiliate principal investigator [PI], oncology physician, Cancer Care Delivery Research [CCDR] Lead) and/or program administrator/supervisor who are willing to be key contacts.
* PRACTICE SITE: Demonstrated support/buy-in from oncology physicians who are willing to enroll patients.
* PRACTICE SITE: Agreement of practice leadership and other individuals at the practice cluster to support/participate in the study activities.
* PRACTICE SITE: If necessary, willingness to participate in a phone interview to determine capacity to implement the ENABLE program.
* INDIVIDUALS AT THE PARTICIPATING PRACTICE: The ENABLE implementation team at each participating practice will include at minimum one ENABLE coach and a coordinator. Other members of the team can include the primary affiliate PI, an oncology physician or investigator, CCDR lead (if different than the coordinator, and/or the program administrator/supervisor) and other professional individuals.
* ONCOLOGY PHYSICIAN: Eligible providers at practices sites are oncology physicians (i.e., medical oncologists or radiation oncologists including trainees) caring for oncology patients. If no oncology physicians are available at the practice, other providers (e.g., advanced practice providers [APPs]) may take on the responsibilities of the oncology physician as laid out in this protocol. We do not require that all physicians at a practice setting agree to participate. Oncology physicians must work at a participating practice cluster with no plans to leave that practice site or retire at the time of enrollment into the study. Physicians (oncologists) may serve in the ENABLE coach role and perform the palliative care assessment, ENABLE sessions and/or monthly follow-up calls per practice discretion if they have completed appropriate training.
* ENABLE COACH: All participating practice clusters will be required to identify one (or more) ENABLE coaches as part of study eligibility to deliver the ENABLE program. The ENABLE coach is responsible for ensuring the ENABLE sessions and follow-up calls are completed per protocol specifications.
* ENABLE COACH: A registered nurse or advanced practice provider (including a nurse practitioner or physician assistant), a physician (e.g., medical and radiation oncologists, including oncology trainees), or other professionals (e.g., social workers, chaplains) with appropriate credentials and experience to deliver ENABLE
* ENABLE COACH: Individuals with an appropriate clinical license (i.e., a registered nurse, advanced practice provider, or physician, as defined above) may perform the palliative care assessment and any ENABLE sessions and follow-up calls the practice chooses to deliver
* ENABLE COACH: Other professionals (e.g., social workers, chaplains) may deliver ENABLE sessions and monthly follow-up calls for which their credentials and experience are appropriate
* ENABLE COACH: ENABLE coaches complete appropriate study training for any content delivered.
* PATIENTS: English-speaking as not all patient measures have been validated in other languages.
* PATIENTS: Age >= 18
* PATIENTS: Willing to complete palliative care assessment and ENABLE sessions.
* PATIENTS: Diagnosed within the last 90 days with an advanced cancer (defined as a newly diagnosed stage III/IV, recurrence, or progressive solid tumor cancer). Patients can receive any cancer treatment for their advanced cancer while participating in this study.

  * The 90-day interval refers to when the patient was made aware of their diagnosis.
* PATIENTS: Expected survival of at least 6 months.
* PATIENTS: Have access to telephone that can receive incoming calls.
* PATIENTS: Able to provide informed consent.

Exclusion Criteria:

* PATIENTS: Received previous palliative care services. (Concurrent palliative care is allowed.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2026-08-23 (Estimated)

PRIMARY OUTCOMES:
Patient completion of the Educate, Nurture, Advise, Before Life Ends (ENABLE) program | Up to 24 weeks
  Defined as having a palliative care assessment and completing at least 4 ENABLE sessions. A logit generalized estimating equation model with exchangeable correlation structure (to account for clustering within practice) will be fitted to a binary patient uptake indicator ("yes" if the patient completed a palliative care assessment and at least 4 ENABLE program sessions and "no" if the patient does not), with the group assignment as the main predictor. Model-predicted uptake proportions, odds ratios, relative risks, and confidence intervals for these measures will be used for interpretation. An additional analysis with sex, group assignment, and an interaction between the two as predictors will be conducted to examine whether this biological variable is a possible moderator of ENABLE program uptake.

SECONDARY OUTCOMES:
Preliminary effectiveness of VLC or TA on patient quality of life and mood outcomes | At 24 weeks
  Will examine and quantify study group differences. A primary analysis, including all patients (either deceased or surviving by the scheduled 24-week follow-up) will be conducted using joint-modeling for longitudinal and time-to-event data to obtain inferences on the longitudinal outcome corrected for non-ignorable missing data due to death. In this approach, submodels for both the longitudinal process and the time-to-event process are estimated simultaneously, with a Cox model for the survival submodel, and a linear mixed-effects model for the longitudinal submodel. The two submodels share random effects for each individual, and these random effects account for both the association between the longitudinal outcome and the risk of death. A sensitivity analysis will also be performed.
Relationship between ENABLE program uptake and patient outcomes | Up to 24 weeks
  Will estimate the relationship between change in patient outcomes (quality of life and mood) using the number of ENABLE sessions completed (ENABLE program uptake) as the main predictor. The crude association between ENABLE sessions and change in patient outcomes will be examined graphically with profile plots, and with linear mixed models to determine whether the relationship is better fitted by a linear, a more complex trend, or as ordinal categorical data. Since the number of ENABLE sessions completed might be dependent on patient characteristics (e.g., sex, illness acuity, age), a covariate adjustment (via an adjusting score) will be conducted on the crude association estimate to determine the change in outcomes attributable to the number of ENABLE sessions completed, above and beyond patient characteristics. The adjusting score will be estimated with a random forest ensemble, based on patient characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Zubkoff, PhD, Principal Investigator — University of Rochester NCORP Research Base
Locations (113):
- United States (113):
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Island Urology-Hilo, Hilo, Hawaii
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Mary's Hospital, Centralia, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center, Springfield, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin

REFERENCES:
- [Derived] Zubkoff L, Lyons KD, Dionne-Odom JN, Hagley G, Pisu M, Azuero A, Flannery M, Taylor R, Carpenter-Song E, Mohile S, Bakitas MA. A cluster randomized controlled trial comparing Virtual Learning Collaborative and Technical Assistance strategies to implement an early palliative care program for patients with advanced cancer and their caregivers: a study protocol. Implement Sci. 2021 Mar 11;16(1):25. doi: 10.1186/s13012-021-01086-3. PMID 33706770